CLINICAL TRIAL: NCT05285488
Title: Impact of Distance Meditation on Non-attachment to the Self and Identity Threat
Acronym: MEDIT-ENLIGNE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-014-MEDIT-ENLIGNE
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Meditation
Keywords: non-attachment to the self; identity threat; meditation; focused attention; contemplation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "focused attention" group (Experimental): adult subjects practicing focused attention meditation
  Interventions: Other: "focused attention" group
- "Contemplation" group (Active Comparator): adult subjects practicing contemplation meditation
  Interventions: Other: "focused attention" group

INTERVENTIONS:
Other: "focused attention" group — "focused attention" group: adult subjects practicing focused attention meditation.
  "contemplation" group: adult subjects practicing contemplation meditation.
  Other Names: "Contemplation" group

SUMMARY:
Meditation is widely recognized for its benefits on both physical and psychological health and more particularly on the prevention of depression relapse. However, despite a lot of literature showing its efficacy, the mechanisms of action underlying its benefits have yet to be specifically identified and empirically tested.

to understand these mechanisms actions, it is essential to distinguish meditative practices. Three different categories of meditation can be distinguished: "Attention Family", "Constructive Family" and "Deconstructive Family" with specific effects for each.

DETAILED DESCRIPTION:
The aim of the study is to compare effects of two types of meditation (focused attention and contemplation) on non-attachment to the self and identity threat.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* aged of 18 and more
* without diagnosed psychiatric pathology
* not practicing meditation
* agreeing to participate in the study

Exclusion Criteria:

- less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
non-attachment to the self | week 6
  Non-attachment to the self evaluated using Adult Self-transcendence Inventory (ASTI).
  ASTI is composed of 10 items. Each item is coded from 1 (totally disagree) to 7 (totally agree) by comparing how they see life at the time of the questionnaire compared to the last 5 years. The overall score ranges from 10 to 70 points.

SECONDARY OUTCOMES:
Identity threat | week 6
  Identity threat evaluated using Cognitive Appraisal Scale (ECP). ECP is composed of 10 items. Each item is coded from 1 (totally disagree) to 6 (totally agree). The overall score ranges from 6 to 60 points

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Reims-Champagne-Ardenne, Reims, Grand Est, France

IPD SHARING:
Plan to Share IPD: No